CLINICAL TRIAL: NCT04527185
Title: Does Endotoxin Administration Increase Alcohol Consumption in Individuals With AUD?
Brief Title: Effect of Endotoxin on Alcohol Consumption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Terril Verplaetse, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000028772; 1R03AA028361-01A1 (NIH)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endotoxin (Experimental): Endotoxin (0.4ng/kg i.v.) will be administered one time during the laboratory session.
  Interventions: Drug: Endotoxin
- Placebo (Placebo Comparator): Administered one time during the laboratory session.
  Interventions: Drug: Endotoxin

INTERVENTIONS:
Drug: Endotoxin — Endotoxin 0.4ng/kg i.v.
  Other Names: Lipopolysaccharide

SUMMARY:
For this protocol, the investigators plan to collect pilot data to examine the effect of endotoxin on drinking behavior in the human laboratory.

DETAILED DESCRIPTION:
This pilot study is a double-blind, placebo-controlled design, which will compare endotoxin (0.4ng/kg i.v.) to placebo (0.0ng/kg) in non-treatment seeking adults meeting criteria for DSM-5 alcohol use disorders (n=32 total, n=16 per group).

Eligibility screening consists of an intake session and a physical exam. Participants meeting eligibility criteria will be randomized to receive a single dose of 0.4ng/kg i.v. endotoxin or placebo during a single laboratory session to evaluate ad-libitum alcohol consumption.

During the laboratory session, endotoxin (or placebo) administration will precede a 2-hour alcohol self-administration period.

Participants will be scheduled for a follow-up appointment to evaluate drinking behavior.

Adverse events are evaluated during the laboratory session and follow-up, and will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65;
2. Able to read and write English;
3. Meets DSM-5 criteria for current (past 6 months) alcohol use disorder;
4. Drinking criteria: Males - Drinks > 14 drinks per week and exceeds 4 drinks per day at least twice per week; Females -Drinks > 7 drinks per week and exceeds 3 drinks per day at least twice per week.
5. Must meet drinking criteria during a consecutive 30-day period within the 90 days prior to baseline;
6. Laboratory sessions will be scheduled such that subjects will not have major responsibilities on the following day which might limit drinking during the self-administration session (e.g., job interview, exam).
7. Negative urine pregnancy test for women.

Exclusion Criteria:

1. Participants with any significant current medical conditions (neurological, cardiovascular [including hypertension or hypotension: sitting BP >160/100 or <90/60mmHg at baseline screening], endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions including HIV;
2. Current DSM-5 substance use disorders, other than alcohol or nicotine;
3. A positive test result at intake appointment on urine drug screens conducted for illicit drugs, excluding cannabis;
4. Past 30 day use of psychoactive drugs including anxiolytics and antidepressants;
5. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD);
6. Suicidal, homicidal or evidence of current (past 6-month) severe mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders;
7. Subjects treatment-seeking or who are currently in treatment for alcohol use;
8. Subjects with medical conditions contraindicating alcohol use (e.g., liver enzymes ≥3× normal);
9. Subjects likely to exhibit clinically significant alcohol withdrawal during the study. We will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments;
10. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current application.
11. Subjects >38 on the Alcohol Use Disorders Identification Test (AUDIT)
12. Subjects with resting pulse >100 at challenge
13. Subjects with recent (past 2 weeks) acute illness or vaccination
14. Subjects with >Grade 2 laboratory abnormalities on screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terril Verplaetse, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomly assigned to endotoxin or placebo prior to the lab session.
Period: Overall Study
Arm/Group | Endotoxin | Placebo
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotoxin | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
Marital Status [Count of Participants; unit: Participants]
  Married | 2 | 0 | 2
  Divorced | 0 | 1 | 1
  Single | 5 | 4 | 9
  Cohabitating | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption
Description: Mean mls of alcohol consumed for endotoxin and placebo groups during 120 minute alcohol self-administration session.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 7 | 6
Milliliters | 37.57 (47.27) | 50.08 (37.58)

ADVERSE EVENTS:
Time Frame: Lab session: +60, +75, +135, +165, +195, +225, +285, +345, +405, +450 minutes following endotoxin administration.
Arm/Group | Endotoxin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Aims on this project were disrupted due to COVID-19 and supplier issues with endotoxin: Clinical research at Yale resumed as of August 1, 2021. Further, there was a significant delay in obtaining endotoxin for use in human subjects. The investigators supply from NIH was depleted and organizing and ordering additional endotoxin from List Laboratories (along with all the regulatory paperwork) took longer than expected. Investigators were without endotoxin from 5/2021 to 1/2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04527185/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04527185/ICF_001.pdf